CLINICAL TRIAL: NCT04758182
Title: Effects of High Intensity Laser Therapy Compared With Ultrasound Therapy on Hemiplegic Shoulder Pain; Randomized Control Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Siriraj Hospital (Other)
Responsible Party: Principal Investigator, Kanyakorn Buspavanich, KANYAKORN BUSPAVANICH M.D., Siriraj Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 053/2563
Record Dates: First submitted 2021-02-15; First posted 2021-02-17 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Hemiplegic Shoulder Pain
MeSH Terms: interventions — Ultrasonic Therapy

STUDY DESIGN:
Intervention Model Description: Double blinded randomize control trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants were blinded; participants in experimental group were received HILT and sham ultrasound, while participants in control group were received ultrasound and sham HILT.
  Outcome assessor was blinded to the treatment group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Experimental group: HILT + sham ultrasound therapy In the experimental group, participants received HILT treatment 1 session per day over a period of 2 consecutive weeks (5 days/week); total 10 sessions. In this study we used HIRO 3.0 device applied to the hemiplegic shoulder and the area of following muscles include upper trapezius, supraspinatus, deltoid, pectoralis minor muscles and the tender points. The treatment consisted of high peak power (3kW), a wavelength of 1064 nm. Two phases of treatment were performed according to Rotator cuff tendinopathy protocol of the device. The total energy administered will be approximately 2500 J. The total treatment time was approximately 10 minutes. They also received sham ultrasound therapy, which performed by applying probe with gel without turning on the device, for 10 minutes.
  Interventions: Device: High intensity laser therapy
- Control group (Active Comparator): Control group: sham HILT + ultrasound therapy In control group, participants received continuous ultrasound therapy for 10 minutes in the same area as an experimental group with Chattanooga intellect mobile ultrasound device. The device was operated at the frequency of 1 MHz, an intensity of 2 W/cm2 and a duty cycle of 100% in the same area of the HILT group. They also received sham HILT, by applying the applicator with pre-recorded sound without starting the device, for 10 minutes. Ultrasound therapy and sham ultrasound were delivered according to the predefined protocol by the physiotherapists.
  Both groups received 3 ROM exercise sessions per day. Participants and their caregiver were educated about proper positioning and manual handling
  Interventions: Device: Ultrasound therapy

INTERVENTIONS:
Device: High intensity laser therapy — Device: HIRO 3.0 device high peak power (3kW), a wavelength of 1064 nm
  Other Names: HILT
  Arms: Experimental group
Device: Ultrasound therapy — Device: Chattanooga intellect mobile ultrasound device frequency of 1 MHz, an intensity of 2 W/cm2 and a duty cycle of 100%
  Arms: Control group

SUMMARY:
Hemiplegic shoulder pain is a common clinical consequence of stroke and can result in significant disability.There are several treatments for Hemiplegic shoulder pain. Patient and family education (ie, range of motion and positioning) is recommended for shoulder pain and shoulder care after stroke, particularly before discharge or transitions in care. Ultrasound therapy is frequently used to relieve pain in hemiplegic shoulder; although there were limited evidences of benefit of ultrasound in hemiplegic shoulder. Laser therapy has become increasing use in hemiplegic shoulder pain. Previous study shows that low level laser therapy significantly reduced pain and improved range of motion in hemiplegic shoulder compared with electrotherapy. High intensity laser therapy (HILT) has been known to reduce pain through multiple pathways including central nervous system pathway, peripheral nervous system pathway and tissues pathway. According to Latest systematic review and meta-analysis, HILT significantly improved pain and disability scores compared with control in musculoskeletal disease especially with neck and back pain. To the best of our knowledge, there is no clinical trial regarding the efficacy of HILT in hemiplegic shoulder pain. Therefore, the aim of our study is to investigate the beneficial effects of HILT on pain reduction, ROM and function in patients with hemiplegic shoulder pain.

DETAILED DESCRIPTION:
Hemiplegic shoulder pain is a common clinical consequence of stroke and can result in significant disability. Shoulder pain can negatively affect rehabilitation outcomes as good shoulder function is a prerequisite for successful transfers, maintaining balance, effective hand function, and performing activities of daily living. The reported prevalence of shoulder pain varies between 5% and 84%, depending on timing and definition of shoulder pain used. An incidence of hemiplegic shoulder pain during the first year range from 1% to 22%. Causes of hemiplegic shoulder pain are multifactorial. Pain is associated with shoulder tissue injury, abnormal joint mechanics, and central nociceptive hypersensitivity. About one third of patients with acute stroke have abnormal ultrasound findings in the hemiplegic shoulder when studied at the time of admission to acute inpatient rehabilitation, including effusion in biceps tendon or subacromial bursa; tendinopathy of biceps, supraspinatus, or subscapularis; and rotator cuff tear There are several treatments for Hemiplegic shoulder pain. Patient and family education (ie, range of motion and positioning) is recommended for shoulder pain and shoulder care after stroke, particularly before discharge or transitions in care. Well- known interventions for Hemiplegic shoulder pain includes botulinum toxin injection, intraarticular steroid injection and transcutaneous electrical nerve stimulation. Nowadays, there are high technology modalities which are less invasive such as ultrasound therapy, extracorporeal shockwave therapy, repetitive transcranial magnetic stimulation and laser therapy.

Ultrasound therapy is frequently used to relieve pain in hemiplegic shoulder; although there were limited evidences of benefit of ultrasound in hemiplegic shoulder. Randomized control trials in 2010 showed that ultrasound therapy significantly reduce pain and increase pain free ROM of post stroke shoulder pain.

However from previous study in1972 showed that ultrasound dose not significantly increases pain free range of motion in the involved shoulders of patients with hemiplegia.

Laser therapy has become increasing use in hemiplegic shoulder pain. Previous study shows that low level laser therapy significantly reduced pain and improved range of motion in hemiplegic shoulder compared with electrotherapy. High intensity laser therapy (HILT) has been known to reduce pain through multiple pathways including central nervous system pathway, peripheral nervous system pathway and tissues pathway. In the central nervous system, laser therapy centrally inhibits pain sensation by increasing the secretion of endogenous opioids such as b-endorphins. In the peripheral nervous system, laser therapy has been reported to decrease the secretion of substance P by peripheral receptors. Laser therapy might increase the latency and decrease the conduction velocity of sensory nerves by inhibiting Aδ- and C-fiber transmission; these in turn may decrease the transmission of pain signals. In tissues, laser therapy may also reduce the release of histamine and bradykinin in injured tissues and increase the pain threshold. HILT increases cell metabolism, vascular permeability, and blood flow in deep tissue structures. Compared to low level laser therapy, HILT have a shorter laser emission time and a longer laser emission interval. Therefore, a large amount of laser irradiation can be delivered to deep tissues.

According to Latest systematic review and meta-analysis, HILT significantly improved pain and disability scores compared with control in musculoskeletal disease especially with neck and back pain. From this study there was insufficient evidence to conclude the efficacy of HILT on shoulder pain. However, in randomized controlled trial which studied the efficacy of HILT in patients with subacromial impingement syndrome showed greater reduction in pain, improvement in articular movement and muscle strength of the affected shoulder after 10 treatment sessions of HILT than did participants receiving Ultrasound therapy over a period of 2 consecutive weeks. In management of frozen shoulder, HILT (3 times per week for 3 weeks) provided significant pain relief at 3 and 8 weeks, but not at the final follow-up time point ( 12 weeks).

To the best of our knowledge, there is no clinical trial regarding the efficacy of HILT in hemiplegic shoulder pain. Therefore, the aim of our study is to investigate the beneficial effects of HILT on pain reduction, ROM and function in patients with hemiplegic shoulder pain.

* Objectives To investigate the beneficial effects of HILT on pain reduction, ROM and function in patients with hemiplegic shoulder pain compared with ultrasound therapy
* Research Process Please specify research procedures, research devices, steps of research process, things that participants/volunteers must do or be treated (such as number of blood drawn, amount of blood drawn, number of appointments, time consuming for participation in the study). If the research proposal is attached, the wordings in Thai and English versions must be the same, including the reference pages in the relevant proposal.

  1. Stroke patients who have hemiplegic shoulder pain and meet with inclusion criteria will be recruited from inpatient department of Department of Rehabilitation Medicine Faculty of Medicine, Siriraj Hospital.
  2. Participants whose characteristics meet the exclusion criteria will be excluded
  3. All participants who are recruited will be provided with an information sheet explaining the study protocol and informed consent.
  4. Sticker determining that the patient was recruited to the shoulder pain research project will be placed in front of patient's chart to inform the practitioner.
  5. The assessor (Physiatrist) will assess participant's baseline demographic data, pain score, affected shoulder range of motion and brunnstrom classification.
  6. After randomization, the participants are divided into 2 groups. Participants will be randomly allocated to experimental group or control group with the help of computer-generated block of four randomization sequence placed in sequentially numbered opaque sealed envelopes by administration staff 6.1 Experimental group: HILT + sham ultrasound therapy participants will receive HILT treatment 1 session per day over a period of 2 consecutive weeks (5 days/week); total 10 sessions.

     In this study the investigators use an HIRO 3.0 device apply to hemiplegic shoulder and the area of following muscles include upper trapezius, supraspinatus, deltoid, pectoralis minor muscles and the tender points.

     The treatment consists of high peak power (3kW), a wave length of 1064 nm. Two phases of treatment will be performed according to Rotator cuff tendinopathy protocol of the device. Two steps are predicted in the initial (fast manual scanning phase) and final (slow scanning phase) phases of the treatment; the intensity used are 810, 970 and 1070 mJ/cm2, respectively. Therefore, the total energy administered will be approximately 2500 J. The total treatment time will be approximately 10 minutes.

     The participants will also receive sham ultrasound therapy for 10 minutes. (HILT and sham HILT will be provided by co-investigator who is a resident of Department of Rehabilitation Medicine Faculty of Medicine, Siriraj Hospital).

     6.2 In control group: sham HILT + ultrasound therapy participants will receive continuous ultrasound therapy for 10 minutes in the same area as an experimental group with Chattanooga intellect mobile ultrasound device. The device will be operated at the frequency of 1 MHz, an intensity of 2 W/cm2 and a duty cycle of 100% in the same area of the HILT group. The participants will also receive sham HILT for 10 minutes. (Ultrasound therapy and sham ultrasound will be provided by Physiotherapists of Department of Rehabilitation Medicine Faculty of Medicine, Siriraj Hospital.)
  7. Both groups will receive 3 ROM exercise sessions per day. First at Physiotherapy gym by the physiotherapists who do ultrasound therapy, second at Occupational therapy room by the occupational therapist and third at bedside by themselves. The researcher who is physiatrist will check for compliance. Participants and their caregiver will be educated about proper positioning and manual handling.
  8. After 10 sessions the assessor who are blind to the intervention groups (Physiatrist) will assess pain score ( numeric rating scale), affected shoulder range of motion with the standard protocol to measure shoulder flexion, abduction, internal and external rotation with goniometer according to the standard text book, brunnstorm classification and side effects.
  9. Participants are permitted to ask for pain killer medication (paracetamol) and pill count will be recorded.

Bobath sling will be worn only while walking, otherwise participants will use pillow support for proper positioning.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. 1st or recurrent stroke onset within 1 year
3. Hemiplegia due to stroke with pain and limited range of motion on the shoulder on the affected side
4. Pain score (Numeric rating scale) ≥ 3
5. Stable medical and neurological conditions
6. Understand Thai.

Exclusion Criteria:

1. Patients with pacemaker
2. Pregnancy
3. Aphasia or could not express their own pain intensity
4. Patients with history of shoulder pain or limited ROM of the affected shoulder prior to stroke onset
5. Patients who had history of trauma or surgery of the shoulder on the affected side
6. Infection or malignancy at the area around affected shoulder
7. central post-stroke pain or complex regional pain syndrome
8. TMSE < 24

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2020-02-27 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain: Numeric rating scale | 2 weeks
  In a Numerical Rating Scale (NRS), patients were asked to circle the number between 0 and 10.
  0 represents 'no pain at all' whereas 10 represents 'the worst pain ever possible. Numerical Rating Scales have shown high correlations with other pain-assessment tools in several studies and it is feasible. In several studies the minimal clinically important difference of NRS is 30%

SECONDARY OUTCOMES:
Shoulder passive range of motion | 2 weeks
  In this study we used the standard protocol to measure shoulder flexion, abduction, internal and external rotation with goniometer according to the standard textbook. The assessor measured each range twice and mean range will be used.
Brunnstrom classification of arm and hand | 2 weeks
  Brunnstrom recovery stage (BRS) is stroke specific and commonly used clinical method to classify the level of post-stroke motor recovery. BRS is a subjective method of classification, and it has also been used as an outcome measure in various studies. It is a reliable, valid, and responsive measuring tool.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine Siriraj hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No